CLINICAL TRIAL: NCT05669651
Title: A Multicenter, Prospective, Randomized Controlled Study to Explore the Efficacy and Safety of Fecal Microbiota Transplantation With Different Bacterial Doses in the Treatment of Recurrent Hepatic Encephalopathy
Brief Title: Explore the Efficacy and Safety of FMT With Different Bacterial Doses in the Treatment of Hepatic Encephalopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hainv Gao (Other)
Responsible Party: Sponsor-Investigator, Hainv Gao, professor, Shulan (Hangzhou) Hospital
Organization: Shulan (Hangzhou) Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Shulan (Hang zhou)2
Record Dates: First submitted 2022-12-14; First posted 2023-01-03 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Hepatic Encephalopathy
Keywords: hepatic encephalopathy; fecal microbiota transplantation
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose of group (Experimental): Complete the fecal bacteria transplantation through the upper digestive tract:
  1. Intestinal preparation: Amoxicillin 0.5g bid, metronidazole 0.4g bid and levofloxacin 0.5g qd for 3 days.
  2. FMT: After 12h of antibiotic discontinuation, the total amount of bacterial liquid was 400ml, 100ml each time, Q12h, 2 days after 12h of antibiotic discontinuation.
  Interventions: Other: Fecal Microbiota Transplantation
- High dose of group (Experimental): Complete the fecal bacteria transplantation through the upper digestive tract:
  1. Intestinal preparation: Amoxicillin 0.5g bid, metronidazole 0.4g bid and levofloxacin 0.5g qd for 3 days.
  2. FMT: After 12h of antibiotic discontinuation, the total amount of bacterial liquid was 800ml, 100ml each time, Q12h, 4 days .
  Interventions: Other: Fecal Microbiota Transplantation

INTERVENTIONS:
Other: Fecal Microbiota Transplantation — Fecal microbiota transplantation (FMT) refers to the transplantation of functional flora from healthy people's feces into patients' intestines to rebuild new intestinal flora and achieve the treatment of intestinal and parenteral diseases. In this study, 100 patients with recurrent hepatic encephalopathy were randomly divided into 1:1 groups to receive FMT with different amounts of bacteria, observe the therapeutic effect and adverse reactions of hepatic encephalopathy, and evaluate the effectiveness and safety of the two groups of patients. At the same time, the blood and stool samples of patients with recurrent hepatic encephalopathy before and after FMT were collected clinically, the composition of bile acid and other metabolites in stool and serum samples was analyzed, and the effective core flora was identified to clarify the mechanism of intestinal bacteria transplantation for the treatment of recurrent hepatic encephalopathy.

SUMMARY:
Hepatic encephalopathy (HE) is one of the most serious complications of end-stage liver disease and an independent predictor of death in patients with liver cirrhosis. Recurrent hepatic encephalopathy is defined as recurrent hepatic encephalopathy after rifaximin combined with lactulose treatment. This project designs a prospective, multicenter cohort study on the treatment of recurrent hepatic encephalopathy with fecal microbiota transplantation, carries out the comparison of fecal microbiota transplantation with different amounts of bacteria, and the dynamic sequencing of the macro genome of the recipient's stool, compares the effectiveness and safety of fecal microbiota transplantation with different amounts of bacteria in the treatment of recurrent hepatic encephalopathy, and explores the internal mechanism of different effects, providing a new idea for the treatment of recurrent HE in clinical practice.

DETAILED DESCRIPTION:
Fecal microbiota transplantation (FMT) refers to the transplantation of functional flora from healthy people's feces into patients' intestines to rebuild new intestinal flora and achieve the treatment of intestinal and parenteral diseases. In this study, 100 patients with recurrent hepatic encephalopathy were randomly divided into 1:1 groups to receive FMT with different amounts of bacteria, observe the therapeutic effect and adverse reactions of hepatic encephalopathy, and evaluate the effectiveness and safety of the two groups of patients. At the same time, the blood and stool samples of patients with recurrent hepatic encephalopathy before and after FMT were collected clinically, the composition of bile acid and other metabolites in stool and serum samples was analyzed, and the effective core flora was identified to clarify the mechanism of intestinal bacteria transplantation for the treatment of recurrent hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old;
2. At least two obvious episodes of hepatic encephalopathy (West-Haven ≥ 2 ) were related to cirrhosis in the first 6 months, and the condition was in remission (West Haven grade 0 or 1) at the time of enrollment. The attack of hepatic encephalopathy caused by gastrointestinal bleeding requiring at least 2 units of blood transfusion, the use of sedatives, renal failure requiring dialysis or central nervous system injury is not recorded as the previous attack;
3. MELD score i ≤ 25 points (score range is 6-40, the higher the score is, the more serious the disease is)
4. Meet the requirements for receiving FMT through nasojejunal tube
5. The subject (or guardian) has signed the informed consent form

Exclusion Criteria:

1. Patients expected to undergo liver transplantation within 1 month
2. Patients with known causes of hepatic encephalopathy (including gastrointestinal bleeding and placement of portal systemic shunt or transjugular intrahepatic portal systemic shunt) within 3 months
3. There are chronic renal insufficiency (creatinine level > 2.0mg/dl), respiratory insufficiency, anemia (HB < 8g / dl), electrolyte abnormalities (serum sodium < 125umol / L; serum calcium > 10mg / dl [2.5umol / l]; or serum potassium < 2.5 mmol / L)
4. Heavy drinking in recent 12 weeks
5. Have used drugs that affect the psychometric score of hepatic encephalopathy (PHEs), such as antidepressants and sedative hypnosis, in recent 4 weeks
6. Patients who are allergic to antibiotics before treatment
7. Infection (pathogen obtained through sterile sites)
8. Patients with chronic endogenous gastrointestinal diseases, such as inflammatory bowel disease (ulcerative colitis, Crohn's disease or microscopic colitis), irritable bowel syndrome
9. Suffering from neurological diseases, such as stroke, epilepsy, dementia and Parkinson's disease
10. Pregnant or lactating patients (urine pregnancy test will be used for examination)
11. Patients who cannot provide informed consent
12. Patients who are unwilling or unable to undergo indwelling nasojejunal tube
13. Other researchers think it is not suitable to be included in this experiment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of the first breakthrough episode of hepatic encephalopathy after FMT. | 12 weeks
  West-Haven Grade ≥2 that occurs within 12 weeks is defined as the first breakthrough episode of hepatic encephalopathy after FMT. Breakthrough attack patients identified as FMT is invalid, no breakthrough attack patients identified as FMT is effective, at the same time compare the advantages and disadvantages of two ways of FMT efficacy.

SECONDARY OUTCOMES:
FMT related serious adverse events | one month
  FMT related serious adverse events
FMT related adverse events | one month
  FMT related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Hainv Gao, doctor, Study Chair — Shulan (Hangzhou) Hospital
Locations (1):
- Shulan (Hangzhou) Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bajaj JS, O'Leary JG, Tandon P, Wong F, Garcia-Tsao G, Kamath PS, Maliakkal B, Biggins SW, Thuluvath PJ, Fallon MB, Subramanian RM, Vargas HE, Lai J, Thacker LR, Reddy KR. Hepatic Encephalopathy Is Associated With Mortality in Patients With Cirrhosis Independent of Other Extrahepatic Organ Failures. Clin Gastroenterol Hepatol. 2017 Apr;15(4):565-574.e4. doi: 10.1016/j.cgh.2016.09.157. Epub 2016 Oct 5. PMID 27720916
- [Result] Bajaj JS, Salzman NH, Acharya C, Sterling RK, White MB, Gavis EA, Fagan A, Hayward M, Holtz ML, Matherly S, Lee H, Osman M, Siddiqui MS, Fuchs M, Puri P, Sikaroodi M, Gillevet PM. Fecal Microbial Transplant Capsules Are Safe in Hepatic Encephalopathy: A Phase 1, Randomized, Placebo-Controlled Trial. Hepatology. 2019 Nov;70(5):1690-1703. doi: 10.1002/hep.30690. Epub 2019 Jun 18. PMID 31038755
- [Result] Butterworth RF. Hepatic Encephalopathy in Cirrhosis: Pathology and Pathophysiology. Drugs. 2019 Feb;79(Suppl 1):17-21. doi: 10.1007/s40265-018-1017-0. PMID 30706423
- [Result] Bajaj JS, Heuman DM, Sanyal AJ, Hylemon PB, Sterling RK, Stravitz RT, Fuchs M, Ridlon JM, Daita K, Monteith P, Noble NA, White MB, Fisher A, Sikaroodi M, Rangwala H, Gillevet PM. Modulation of the metabiome by rifaximin in patients with cirrhosis and minimal hepatic encephalopathy. PLoS One. 2013;8(4):e60042. doi: 10.1371/journal.pone.0060042. Epub 2013 Apr 2. PMID 23565181
- [Result] McDonald LC, Gerding DN, Johnson S, Bakken JS, Carroll KC, Coffin SE, Dubberke ER, Garey KW, Gould CV, Kelly C, Loo V, Shaklee Sammons J, Sandora TJ, Wilcox MH. Clinical Practice Guidelines for Clostridium difficile Infection in Adults and Children: 2017 Update by the Infectious Diseases Society of America (IDSA) and Society for Healthcare Epidemiology of America (SHEA). Clin Infect Dis. 2018 Mar 19;66(7):e1-e48. doi: 10.1093/cid/cix1085. PMID 29462280
- [Result] Zhang F, Cui B, He X, Nie Y, Wu K, Fan D; FMT-standardization Study Group. Microbiota transplantation: concept, methodology and strategy for its modernization. Protein Cell. 2018 May;9(5):462-473. doi: 10.1007/s13238-018-0541-8. Epub 2018 Apr 24. PMID 29691757
- [Result] DuPont HL. Review article: the antimicrobial effects of rifaximin on the gut microbiota. Aliment Pharmacol Ther. 2016 Jan;43 Suppl 1:3-10. doi: 10.1111/apt.13434. PMID 26618921
- [Result] Vrieze A, Van Nood E, Holleman F, Salojarvi J, Kootte RS, Bartelsman JF, Dallinga-Thie GM, Ackermans MT, Serlie MJ, Oozeer R, Derrien M, Druesne A, Van Hylckama Vlieg JE, Bloks VW, Groen AK, Heilig HG, Zoetendal EG, Stroes ES, de Vos WM, Hoekstra JB, Nieuwdorp M. Transfer of intestinal microbiota from lean donors increases insulin sensitivity in individuals with metabolic syndrome. Gastroenterology. 2012 Oct;143(4):913-6.e7. doi: 10.1053/j.gastro.2012.06.031. Epub 2012 Jun 20. PMID 22728514
- [Result] Moayyedi P, Surette MG, Kim PT, Libertucci J, Wolfe M, Onischi C, Armstrong D, Marshall JK, Kassam Z, Reinisch W, Lee CH. Fecal Microbiota Transplantation Induces Remission in Patients With Active Ulcerative Colitis in a Randomized Controlled Trial. Gastroenterology. 2015 Jul;149(1):102-109.e6. doi: 10.1053/j.gastro.2015.04.001. Epub 2015 Apr 7. PMID 25857665
- [Result] Sender R, Fuchs S, Milo R. Are We Really Vastly Outnumbered? Revisiting the Ratio of Bacterial to Host Cells in Humans. Cell. 2016 Jan 28;164(3):337-40. doi: 10.1016/j.cell.2016.01.013. PMID 26824647
- [Result] Olson MA, Cuff L. Molecular docking of superantigens with class II major histocompatibility complex proteins. J Mol Recognit. 1997 Nov-Dec;10(6):277-89. doi: 10.1002/(SICI)1099-1352(199711/12)10:63.0.CO;2-X. PMID 9770652
- [Result] Human Microbiome Project Consortium. Structure, function and diversity of the healthy human microbiome. Nature. 2012 Jun 13;486(7402):207-14. doi: 10.1038/nature11234. PMID 22699609
- [Result] Qin J, Li R, Raes J, Arumugam M, Burgdorf KS, Manichanh C, Nielsen T, Pons N, Levenez F, Yamada T, Mende DR, Li J, Xu J, Li S, Li D, Cao J, Wang B, Liang H, Zheng H, Xie Y, Tap J, Lepage P, Bertalan M, Batto JM, Hansen T, Le Paslier D, Linneberg A, Nielsen HB, Pelletier E, Renault P, Sicheritz-Ponten T, Turner K, Zhu H, Yu C, Li S, Jian M, Zhou Y, Li Y, Zhang X, Li S, Qin N, Yang H, Wang J, Brunak S, Dore J, Guarner F, Kristiansen K, Pedersen O, Parkhill J, Weissenbach J; MetaHIT Consortium; Bork P, Ehrlich SD, Wang J. A human gut microbial gene catalogue established by metagenomic sequencing. Nature. 2010 Mar 4;464(7285):59-65. doi: 10.1038/nature08821. PMID 20203603
- [Derived] Zou P, Bi Y, Tong Z, Wu T, Li Q, Wang K, Fan Y, Zhao D, Wang X, Shao H, Huang H, Ma S, Qian Y, Zhang G, Liu X, Jin Q, Ru Q, Qian Z, Sun W, Chen Q, You L, Wang F, Zhang X, Qiu Z, Lin Q, Lv J, Zhang Y, Geng J, Mao R, Liu J, Zheng Y, Ding F, Wang H, Gao H. Comparisons of efficacy and safety of 400 or 800 ml bacterial count fecal microbiota transplantation in the treatment of recurrent hepatic encephalopathy: a multicenter prospective randomized controlled trial in China. Trials. 2024 Nov 27;25(1):799. doi: 10.1186/s13063-024-08578-9. PMID 39605077